CLINICAL TRIAL: NCT05684068
Title: Dimensional Changes of Autogenous Free Epithelialized Gingival Grafts on Different Bed Preparations Among Dental Patients With Thin Tissue Phenotypes: A Randomized Clinical Trial
Brief Title: Dimensional Changes: Randomized Clinical Trial
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Iowa (Other)
Responsible Party: Principal Investigator, Carlos Garaicoa Pazmino, Clinical Assistant Professor, University of Iowa
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 202207368
Record Dates: First submitted 2023-01-04; First posted 2023-01-13 (Actual); Last update posted 2025-08-19 (Actual); Status verified 2025-08

CONDITIONS: Gingival Recession
MeSH Terms: conditions — Gingival Recession

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Gum Graft Placed on Denuded Bone (Experimental): Subjects in this arm will have a free epithelialized gingival/mucosal graft (gum graft) placed on full thickness periosteal bed preparation where all of the tissue was removed (test group).
  Interventions: Procedure: Gum Graft Placed on Denuded Bone
- Gum Graft Placed on Split Thickness Periosteal Bed Preparation (Active Comparator): Group B will have a free epithelialized gingival/mucosal graft (gum graft) on split thickness periosteal bed preparation where only a portion of the tissue was removed (control group).
  Interventions: Procedure: Gum Graft Placed on Split Thickness Periosteal Bed Preparation

INTERVENTIONS:
Procedure: Gum Graft Placed on Denuded Bone — The provider will administer local anesthesia into the subject's gum in order to numb both the subject's donor and recipient areas for gum grafts. Next, the provider will use a surgical blade to dissect the gum graft from the subject's donor site. At the subject's recipient gum recession defect site, the provider will remove all of the subject's tissue, so that the bone is fully exposed before placing a gum graft from the donor site. Afterward, the provider will place sutures in the subject's recipient site in order to promote healing/re-growth.
  Arms: Gum Graft Placed on Denuded Bone
Procedure: Gum Graft Placed on Split Thickness Periosteal Bed Preparation — The provider will administer local anesthesia into the subject's gum in order to numb both the subject's donor and recipient areas for gum grafts. Next, the provider will use a surgical blade to dissect the gum graft from the subject's donor site. At the subject's recipient gum recession defect site, the provider will dissect some of the tissue at the subject's recipient site but still keep a small layer of tissue at the subject's recipient site before placing a gum graft from the donor site. Afterward, the provider will place sutures in the subject's recipient site in order to promote healing/re-growth.
  Arms: Gum Graft Placed on Split Thickness Periosteal Bed Preparation

SUMMARY:
The goal of this clinical trial is to evaluate the dimensional changes in the short and long-term in patients with thin gum tissues who have gum grafts placed on either denuded bone or gum grafts placed on a bone with some tissues remaining.

The main question this study aims to answer is:

- Does the placement of free-epithelized gingival grafts (gum grafts) on full thickness bed preparation (having all of the tissue removed from the bone) lead to similar clinical, digital, and patient-related outcomes and measurements over a period of 12 months versus split thickness bed preparation (where a small layer of tissue is left over the bone) in patients with thin gum tissue phenotypes (gum tissue is generally less than 1.5 millimeters) who are in need of soft tissue augmentation procedures?

Participants will be asked to attend 8 visits, which include: (i) screening visit, (ii) prophylaxis visit, (iii) random assignment to Group A or Group B along with surgery and digital data collection, (iv) 2-week post-operative visit, (v) 6-week post-operative visit, (vi) 3-month follow-up visit, (vii) 6-month follow-up visit, (viii) 12-month follow-up visit. Also, Group A will have a free epithelialized gingival/mucosal graft (gum graft) placed on full thickness periosteal bed preparation where all of the tissue was removed (test group). Group B will have a free epithelialized gingival/mucosal graft (gum graft) on split thickness periosteal bed preparation where only a portion of the tissue was removed (control group). Researchers will compare Group A and Group B to see if there is a difference in clinical, digital, and patient-related outcomes and measurements over a period of 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Patients 18-95 years of age
* Inactive periodontal disease
* Lack of, or an insufficient (less than 2 millimeters) band of keratinized tissue width on the buccal site (closest to the cheek)
* Shallow vestibule depth (the space between the soft tissue (lips and cheeks), and the teeth and gums)
* Thin gingival phenotype (less than 1.5mm of gum tissue depth).
* Aberrant frenum attachment in need of free-epithelized gingival grafts.
* At least one RT1, 2, or 3 (Cairo's classification) gingival recession defect on the mandibular anterior sextant (Teeth #22-27).
* Non-smokers or past smokers (those who have stopped at minimum 6 months ago).
* Patient willing and able to follow instruction related to the study procedures.

Exclusion Criteria:

* Previous soft tissue augmentation procedures at the area of interest.
* Current smokers (Light smokers meaning less than 10 cigarettes/day, heavy smokers meaning more than 10 cigarettes/day, or social smokers)
* Uncontrolled systemic disease (uncontrolled diabetes defined by blood sugar HbA1c greater than 7%)
* Any active local or systemic infections
* Any diseases or medications that may compromise normal wound healing
* Currently receiving chemotherapy or radiotherapy or a history of radiotherapy in head and neck area.
* Severe hematologic (blood) disorders
* Pregnancy or nursing mother
* Patients undergoing orthodontic therapy
* Patients taking antibiotics in the past 3 months

Ages: 18 Years to 95 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2028-08 (Estimated); Primary Completion 2030-07 (Estimated); Study Completion 2031-03 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline in Gingival Thickness as assessed by measurement. | Multiple time points (i.e., Baseline, 3 months, 6 months, 12 months)
  Tissue changes will be assessed in millimeters and percentage.

CONTACTS AND LOCATIONS:
Overall Officials: Carlos Garaicoa, DDS, MS, Principal Investigator — University of Iowa College of Dentistry
Locations (1):
- University of Iowa College of Dentistry and Dental Clinics, Iowa City, Iowa, United States

IPD SHARING:
Plan to Share IPD: No